CLINICAL TRIAL: NCT03267537
Title: Non-inferiority Study of Telemedicine Versus Conventional CBT-I in Recently Hospitalized Patients With Insomnia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Arizona (Other)
Collaborators: American Academy of Sleep Medicine (Other)
Responsible Party: Principal Investigator, Sairam Parthasarathy, Professor of Medicine, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1545864655443n/a
Record Dates: First submitted 2017-06-14; First posted 2017-08-30 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Insomnia
Keywords: Insomnia; Sleep; Telemedicine
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Observers will be blinded to subjects group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional office-based CBT-I (Active Comparator): CBT-I will be delivered by a licensed clinical psychologist in weekly sessions lasting up to 1 hour. There will be 6 CBT-I sessions over the course of therapy with the option of an additional 2 treatments if deemed necessary by the clinical psychologist.
  Interventions: Behavioral: Conventional office-based CBT-I
- Telemedicine based CBT-I (Experimental): The treatment will be the exact same as the active comparator group, with the same clinical psychologist doing the office-based CBT-I, but will be administered through a telemedicine modality
  Interventions: Behavioral: Telemedicine CBT-I

INTERVENTIONS:
Behavioral: Telemedicine CBT-I — Will be administered in a manner similar to the conventional CBT-I arm except that the patient would not be required to make office visits
  Arms: Telemedicine based CBT-I
Behavioral: Conventional office-based CBT-I — Conventional office-based CBT-I
  Arms: Conventional office-based CBT-I

SUMMARY:
Insomnia is a common medical condition that has a deleterious effect on emotional status, health-related quality of life, and has been associated with hospitalizations and all-cause mortality. Recently hospitalized patients who are recuperating in their homes would find it difficult to return for weekly visits with a clinical psychologist and therefore could benefit from the convenience of CBT-I treatment administered in the comfort of their homes via the wireless iPAD and video chat software. In patients who are recently discharged from the hospital, we wish to assess whether telemedicine-based CBT-I is comparable to conventional office-based CBT-I in the efficacy for treating insomnia. Research aiming to improve understanding of whether insomnia represents a modifiable risk factor for re-hospitalizations in patients who are high utilizers of healthcare services is an important area of future research.

DETAILED DESCRIPTION:
Insomnia is a common and distressing medical condition that affects nearly 20% of U.S. adults, and persistent (or chronic) insomnia affects nearly 10-15% of U.S. adults. In a community-based prospective observational study, preliminary data suggests that insomnia is associated with hospitalizations due to cardiovascular, cancer, or any cause over a 4-year period. Cognitive Behavioral Therapy for Insomnia (CBT-I) is considered the gold-standard in the treatment of insomnia. There are 5 components of CBT-I, sleep restriction therapy, stimulus control instructions, relaxation training, cognitive therapy, and sleep hygiene education. In an ongoing study of CBT-I in recently hospitalized patients, the investigators found a high prevalence of insomnia (80%) and were able to administer CBT-I in the participants' home via iPADs with wireless connectivity and secure video-chat software. Recently hospitalized patients who are recuperating in their homes would find it difficult to return for weekly visits with a clinical psychologist and therefore could benefit from the convenience of CBT-I treatment administered in the patient's homes via the wireless iPAD and video chat software. The AASM SleepTM platform could conceivably allow performance of CBT-I without the added expense of an iPAD. The investigators are proposing to perform a non-inferiority trial of telemedicine CBT-I (AASM SleepTM) versus conventional office-based CBT-I that is performed in patients with insomnia who have been recently discharged from the hospital. The investigators will measure the following outcomes: insomnia severity index (primary outcome) and patient satisfaction. In the future, the investigators' program of research aims to improve understanding of whether insomnia represents a modifiable risk factor for re-hospitalizations in patients who are high utilizers of healthcare services.

Specific Aim 1: To perform comparative effectiveness research of CBT-I administered by telemedicine versus conventional office-based CBT-I on insomnia severity in recently hospitalized patients.

Hypothesis #1: In recently hospitalized patients with insomnia, after six weeks of CBT-I treatment, the mean improvement in ISI score among patients treated by telemedicine CBT-I (AASM SleepTM) would be no more than 3-points less than that in patients treated by conventional office-based CBT-I.

Specific Aim 2: To perform comparative effectiveness research of CBT-I administered by telemedicine versus conventional office-based CBT-I on patient satisfaction.

Hypothesis #2: In recently hospitalized patients with insomnia, after six weeks of CBT-I treatment, the mean improvement in patient satisfaction score (Consumer Assessment of Health Plans Survey [CAHPS v4.0] item) among patients treated by telemedicine CBT-I (AASM SleepTM) would be no more than 1-point less than that in patients treated by conventional office-based CBT-I.

ELIGIBILITY:
Inclusion Criteria:

* Medically ill patients with recent hospitalization who are being discharged to home.
* ISI score of > 10 (chronic insomnia)
* Age > 18 years
* Ability to provide informed consent
* Willingness to undergo sleep study

Exclusion Criteria:

* Presence of untreated sleep disorder that requires treatment independent of insomnia (Narcolepsy, restless leg syndrome, or REM sleep behavior disorder)
* Patients with severe debilitating neurological disease (end-stage Alzheimer's, large stroke, or other debilitating neurological disease) or any other condition that renders patients incapable of providing informed consent
* History of Bipolar disease; current or past (< 6 months) history of suicidality or suicidal ideation
* Active substance abuse or alcoholism
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2017-06-13 (Actual); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Baseline and after receiving CBT-I (~6 weeks)
  A 7-item questionnaire used to assess insomnia severity with a score ranging between 0 to 28. Each questionnaire item addresses an aspect about sleep that is rated by the respondent on a 5-point scale (i.e., 0=no problem & 4=very severe problem) Change in ISI score will be assessed between baseline and following CBT-I treatment over a 6 week period.

SECONDARY OUTCOMES:
Consumer Assessment of Health Plans Survey (CAHPS v4.0) item | Administered at baseline and at the end of receiving CBT-I (~6 weeks)
  Health plan member's satisfaction with care on 0 to 10 scale (0 is the "worst " and 10 is the "best health plan possible"). Change in CAHPS score will be measured

OTHER OUTCOMES:
Wake After Sleep Onset (WASO) | Sleep diaries are completed daily and actiwatch is worn continuously during the treatment period (~6 weeks)
  WASO is defined as the number of minutes spent awake after sleep onset. This is going to be measured by wrist actigraphy and sleep diaries. Change in WASO will be assessed over the intervention period
Sleep Onset Latency (SOL) | Sleep diaries are completed daily and actiwatch is worn continuously during the treatment period (~6 weeks)
  SOL is the number of minutes that it takes to fall asleep. This is going to be measured by wrist actigraphy and sleep diaries. Change in SOL will be assessed over the intervention period
Pittsburgh Sleep Quality Index (PSQI) | Administered at baseline and at the end of receiving CBT-I (~6 weeks)
  Provides a subjective assessment of sleep quality. Change in PSQI score will be assessed between baseline and 6-week follow-up.
SF-36 Health Survey | Administered at baseline, at the end of receiving CBT-I (~6 weeks), at 2 weeks following treatment, and at 12 weeks following treatment
  A 36 item health status assessment tool, which measures general health and quality of life. Change in various dimensions of the SF-36 will be assessed over the 6-week period.
Re-hospitalizations | Administered at the time of hospital discharge and at the end of receiving CBT-I (~6 weeks)
  Composite number of hospital readmissions over 6 weeks.
Healthcare utilization | Administered at the time of hospital discharge and at the end of receiving CBT-I (~6 weeks)
  Composite number of visits to any of the following locations of healthcare service for care delivery: Emergency room, urgent care, as well as unscheduled and scheduled clinic visits.
Epworth Sleepiness Scale (ESS) | Administered at baseline and at the end of receiving CBT-I (~6 weeks)
  A measure of sleepiness. Change in ESS score will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona (Banner University Medical Center - Tucson & Banner University Medical Center - South), Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buysse DJ. Insomnia. JAMA. 2013 Feb 20;309(7):706-16. doi: 10.1001/jama.2013.193. PMID 23423416
- [Background] Kyle SD, Morgan K, Espie CA. Insomnia and health-related quality of life. Sleep Med Rev. 2010 Feb;14(1):69-82. doi: 10.1016/j.smrv.2009.07.004. Epub 2009 Dec 4. PMID 19962922
- [Background] Parthasarathy S, Vasquez MM, Halonen M, Bootzin R, Quan SF, Martinez FD, Guerra S. Persistent insomnia is associated with mortality risk. Am J Med. 2015 Mar;128(3):268-75.e2. doi: 10.1016/j.amjmed.2014.10.015. Epub 2014 Oct 16. PMID 25447616
- [Background] Foley DJ, Monjan AA, Brown SL, Simonsick EM, Wallace RB, Blazer DG. Sleep complaints among elderly persons: an epidemiologic study of three communities. Sleep. 1995 Jul;18(6):425-32. doi: 10.1093/sleep/18.6.425. PMID 7481413
- [Background] Althuis MD, Fredman L, Langenberg PW, Magaziner J. The relationship between insomnia and mortality among community-dwelling older women. J Am Geriatr Soc. 1998 Oct;46(10):1270-3. doi: 10.1111/j.1532-5415.1998.tb04544.x. PMID 9777910
- [Background] Newman AB, Spiekerman CF, Enright P, Lefkowitz D, Manolio T, Reynolds CF, Robbins J. Daytime sleepiness predicts mortality and cardiovascular disease in older adults. The Cardiovascular Health Study Research Group. J Am Geriatr Soc. 2000 Feb;48(2):115-23. doi: 10.1111/j.1532-5415.2000.tb03901.x. PMID 10682939
- [Background] Rockwood K, Davis HS, Merry HR, MacKnight C, McDowell I. Sleep disturbances and mortality: results from the Canadian Study of Health and Aging. J Am Geriatr Soc. 2001 May;49(5):639-41. doi: 10.1046/j.1532-5415.2001.49125.x. PMID 11380758
- [Background] Nilsson PM, Nilsson JA, Hedblad B, Berglund G. Sleep disturbance in association with elevated pulse rate for prediction of mortality--consequences of mental strain? J Intern Med. 2001 Dec;250(6):521-9. doi: 10.1046/j.1365-2796.2001.00913.x. PMID 11902821
- [Background] Mallon L, Broman JE, Hetta J. Sleep complaints predict coronary artery disease mortality in males: a 12-year follow-up study of a middle-aged Swedish population. J Intern Med. 2002 Mar;251(3):207-16. doi: 10.1046/j.1365-2796.2002.00941.x. PMID 11886479
- [Background] Suzuki E, Yorifuji T, Ueshima K, Takao S, Sugiyama M, Ohta T, Ishikawa-Takata K, Doi H. Sleep duration, sleep quality and cardiovascular disease mortality among the elderly: a population-based cohort study. Prev Med. 2009 Aug-Sep;49(2-3):135-41. doi: 10.1016/j.ypmed.2009.06.016. Epub 2009 Jun 30. PMID 19573557
- [Background] Rod NH, Vahtera J, Westerlund H, Kivimaki M, Zins M, Goldberg M, Lange T. Sleep disturbances and cause-specific mortality: Results from the GAZEL cohort study. Am J Epidemiol. 2011 Feb 1;173(3):300-9. doi: 10.1093/aje/kwq371. Epub 2010 Dec 30. PMID 21193534
- [Background] Almeida OP, Alfonso H, Yeap BB, Hankey G, Flicker L. Complaints of difficulty to fall asleep increase the risk of depression in later life: the health in men study. J Affect Disord. 2011 Nov;134(1-3):208-16. doi: 10.1016/j.jad.2011.05.045. Epub 2011 Jun 15. PMID 21680026
- [Background] Eaker ED, Pinsky J, Castelli WP. Myocardial infarction and coronary death among women: psychosocial predictors from a 20-year follow-up of women in the Framingham Study. Am J Epidemiol. 1992 Apr 15;135(8):854-64. doi: 10.1093/oxfordjournals.aje.a116381. PMID 1585898
- [Background] Vgontzas AN, Liao D, Pejovic S, Calhoun S, Karataraki M, Basta M, Fernandez-Mendoza J, Bixler EO. Insomnia with short sleep duration and mortality: the Penn State cohort. Sleep. 2010 Sep;33(9):1159-64. doi: 10.1093/sleep/33.9.1159. PMID 20857861
- [Background] Li Y, Zhang X, Winkelman JW, Redline S, Hu FB, Stampfer M, Ma J, Gao X. Association between insomnia symptoms and mortality: a prospective study of U.S. men. Circulation. 2014 Feb 18;129(7):737-46. doi: 10.1161/CIRCULATIONAHA.113.004500. Epub 2013 Nov 13. PMID 24226807
- [Background] Haynes PL, Parthasarathy S, Kersh B, Bootzin RR. Examination of insomnia and insomnia treatment in psychiatric inpatients. Int J Ment Health Nurs. 2011 Apr;20(2):130-6. doi: 10.1111/j.1447-0349.2010.00711.x. PMID 21371228
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Schmittdiel J, Mosen DM, Glasgow RE, Hibbard J, Remmers C, Bellows J. Patient Assessment of Chronic Illness Care (PACIC) and improved patient-centered outcomes for chronic conditions. J Gen Intern Med. 2008 Jan;23(1):77-80. doi: 10.1007/s11606-007-0452-5. Epub 2007 Nov 21. PMID 18030539
- [Background] Michelson D, Snyder E, Paradis E, Chengan-Liu M, Snavely DB, Hutzelmann J, Walsh JK, Krystal AD, Benca RM, Cohn M, Lines C, Roth T, Herring WJ. Safety and efficacy of suvorexant during 1-year treatment of insomnia with subsequent abrupt treatment discontinuation: a phase 3 randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2014 May;13(5):461-71. doi: 10.1016/S1474-4422(14)70053-5. Epub 2014 Mar 27. PMID 24680372
- [Background] Morin CM, Vallieres A, Guay B, Ivers H, Savard J, Merette C, Bastien C, Baillargeon L. Cognitive behavioral therapy, singly and combined with medication, for persistent insomnia: a randomized controlled trial. JAMA. 2009 May 20;301(19):2005-15. doi: 10.1001/jama.2009.682. PMID 19454639
- [Background] Buysse DJ, Ancoli-Israel S, Edinger JD, Lichstein KL, Morin CM. Recommendations for a standard research assessment of insomnia. Sleep. 2006 Sep;29(9):1155-73. doi: 10.1093/sleep/29.9.1155. PMID 17040003